CLINICAL TRIAL: NCT03667989
Title: Single-photon Emission Computed Tomography for Prediction and Evaluation of Cardiac Resynchronization Therapy Efficacy in Chronic Heart Failure Patients
Brief Title: SPECT-based Prediction and Evaluation of CRT Efficacy in CHF
Acronym: MIBGinCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIBGinCRT
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2019-09

CONDITIONS: Chronic Heart Failure
Keywords: SPECT; 123I-MIBG; Chronic heart failure; Cardiac resynchronization therapy; CZT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 123I-MIBG CZT SPECT (Other): Patients with ischemic and non-ischemic heart failure with indications for CRT. Assessment of cardiac sympathetic innervation by 123IMIBG CZT SPECT.
  Interventions: Diagnostic Test: Assessment of cardiac sympathetic innervation by 123I-MIBG

INTERVENTIONS:
Diagnostic Test: Assessment of cardiac sympathetic innervation by 123I-MIBG — Assessment of cardiac sympathetic innervation by 123I-MIBG CZT SPECT

SUMMARY:
This study evaluates the state of the cardiac sympathetic activity and the severity of ventricular dyssynchrony in chronic heart failure patients and assesses the capabilities of radionuclide indication methods in determining the prognosis and evaluating the results of cardiac resynchronization therapy in chronic heart failure patients.

DETAILED DESCRIPTION:
In heart failure, abnormal activation of cardiac sympathetic system has been shown to be of pathophysiological significance. However, the left ventricular (LV) dyssynchrony has a detrimental effect on LV systolic and diastolic functions in heart failure patients. The effects of LV dyssynchrony on cardiac sympathetic activity are not yet fully understood. Dilated cardiomyopathy is a common cause of severe chronic heart failure. Cardiac resynchronization therapy (CRT) is a disease modifying device-driven treatment that can reduce morbidity and mortality in patients with heart failure. However, this type of treatment does not lead to the expected results in 25% to 30% of patients despite the successful implantation of a CRT device. In addition, CRT is associated with high cost and potential morbidity. Therefore, the search for new highly informative criteria for selecting patients for this type of treatment remains a relevant task of modern medicine. It is expected that the results obtained will complement and expand current state of knowledge regarding the relationships between cardiac remodeling processes and the state of cardiac sympathetic activity. In addition, obtained data will allow to predict LV remodeling dynamics after the correction of contractile dysfunction of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure NYHA III and IV class
* LVEF ≤ 35 %
* QRS ≥ 150 ms on ECG
* The presence of LBBB on ECG
* Sinus rhythm
* Optimal pharmacological treatment of heart failure

Exclusion Criteria:

* Contraindications to SPECT due to hypersensitivity to radiopharmacuticals such as 2-methoxy-isobutyl-isonitrile-(99mTc) and (123)I-Meta-iodobenzylguanidine or any of the excipients
* Pregnancy
* Breastfeeding
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
CRT response | One year
  ESV decreasing equal or more than 15%

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Popov, MD, PhD, Study Director — Tomsk NRMC
Locations (1):
- Cardiology Research Institute, Tomsk NRMC, Tomsk, Tomsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atabekov T, Korepanov V, Krivolapov S, Khlynin M, Afanasiev S, Golubenko M, Batalov R, Popov S. Mitochondrial DNA Polymorphisms of Peripheral Blood Mononuclear Cells Associated with Sustained Ventricular Tachycardia in Patients with Cardioverter-Defibrillator Implantation Indications. Rev Cardiovasc Med. 2025 Mar 17;26(3):26744. doi: 10.31083/RCM26744. eCollection 2025 Mar. PMID 40160580